CLINICAL TRIAL: NCT02997670
Title: Quartet Lead With Defibrillator Multisite Algorithmic Cardiac Resynchronisation Therapy Optimisation
Acronym: QUARTRMASTER
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Work focused in other areas, other groups working on this.
Sponsor: Cardiff and Vale University Health Board (Other Government)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Freya Lodge, Clinical Research Fellow, Cardiff and Vale University Health Board
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16/WA/0370 186610
Record Dates: First submitted 2016-12-07; First posted 2016-12-20 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure, Systolic
Keywords: Cardiac resynchronization pacing therapy
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main patient cohort (Experimental): Algorithmic Cardiac Resynchronisation Therapy Optimisation; Patients requiring CRT-D enrolled to receive algorithmic CRT optimisation at their device implantation. They will then be programmed to standard CRT settings for 12 weeks. Assessments will be performed and they will again undergo CRT optimisation using the specified algorithm. This time, they will be programmed to the settings giving maximal cardiac output on echocardiography, as assessed by LVOT VTI. After a further 12 weeks, they will again undergo assessment and the study will terminate.
  Interventions: Other: Algorithmic Cardiac Resynchronisation Therapy Optimisation

INTERVENTIONS:
Other: Algorithmic Cardiac Resynchronisation Therapy Optimisation — Use of a computer algorithm to run through multiple combinations of pacing options in patients who have a Cardiac resynchronisation pacemaker with defibrillator where a quadripolar lead has been implanted. These quadripolar leads offer extra options for pacing locations across the heart, as well as for different combinations and sequences of pacing stimuli.

SUMMARY:
Cardiac resynchronisation therapy (CRT) improves outcomes and symptoms in selected patients with heart failure. However, around one third of suitable patients do not demonstrate benefit following device implantation when assessed by echocardiography (heart scanning). This group has poorer outcomes.

Response rate can be enhanced by altering timing delays between the pacing leads, but some patients still fail to improve.

Quadripolar left ventricular leads are now widely used in CRT. The lead's four poles increase the number of conformations available to the programmer, allowing multiple vectors to be programmed simultaneously or sequentially. This allows programming to avoid, for example, a patch of scar and find an area that will respond better to pacing. This technique is known as multi-site pacing. CRT is often implanted along with a defibrillator lead in the right ventricle, known as CRT-D. The defibrillator lead offers further combinations for pacing.

Goal of Research To evaluate an algorithm for assessing different multi-site pacing combinations in optimisation of CRT

Outline The investigators will recruit 24 consecutive patients undergoing CRT-D implantation for conventional indications at our hospital. At baseline, patients will undergo echocardiography, exercise testing and assessments of functional ability and quality of life. The device will be implanted as standard. Optimisation will be performed with an algorithm using different vector combinations and assessing the heart's efficiency through echocardiography and invasive pressure monitoring. The pacemaker will be programmed with standard settings. After twelve weeks, the baseline investigations and optimisation algorithm will be repeated and the device programmed according to the maximum efficiency. After a further 12 weeks, the same parameters will be measured to look for improved response to CRT.

Potential Benefit To increase the response rate to cardiac resynchronisation therapy and improve reliability of the technique

DETAILED DESCRIPTION:
Study Design: This is an open-label, single centre, prospective, cohort study to assess the effect of algorithmic, echocardiography-guided optimisation of CRT-D following implantation of a left ventricular quadripolar lead.

Introduction and background:

There is now considerable evidence that cardiac resynchronisation therapy (CRT) improves outcomes and symptoms in patients with heart failure. However, around a third of patients do not demonstrate any haemodynamic or functional benefit following device implantation. Earlier studies have used a cut-off of 15% reduction in left ventricular end-systolic volume to define response to CRT.

Failure to respond to CRT is felt to be multifactorial. Issues include:

* Anatomical limitations in terms of lead placement (the lead must be placed within a branch of the coronary sinus vein and therefore targeting to the site of maximum contraction delay can be difficult)
* Presence of areas of scar tissue, which are resistant to being paced
* Phrenic nerve stimulation with some pacing sites. The phrenic nerve runs close to the heart and may be stimulated by the pacemaker, with the effect that the patient's diaphragm is stimulated and they experience persistent hiccups.
* High pacing thresholds, which means that increased power from the pacemaker must be used to create a successful pacing stimulus (capture) and that in some instances, capture may not be achieved. This can be due to scar or to poor contact with the heart tissue.

Previous work has demonstrated that response can be improved in some patients by optimisation of inter- and intra-ventricular dyssynchrony and atrio-ventricular delay. However, this optimisation is limited by the fixed location of the leads after implantation, with pacing possible from the lead tip only. Multi-site pacing (MSP) with a quadripolar left ventricular lead has been introduced to increase the number of conformations available to the programmer and is especially useful in reducing phrenic nerve capture. Additionally, multiple vectors can be programmed sequentially or simultaneously, allowing for incorporation of a greater number of myocardial segments. Quadripolar left ventricular leads are now being routinely used in many hospitals. They offer new opportunities for optimising CRT-D (resynchronisation-defibrillator) devices by altering the pacing vectors between the four different poles on the lead and the two defibrillator coils to give hundreds of possible pacing combinations.

Several recent studies have been published looking at the effect of multi-site pacing on effectiveness of CRT therapy. Generally these employ limited vector combinations, but have already demonstrated beneficial effects on haemodynamics and echocardiographic measures of heart function. The evaluation of an algorithm that examines many more vector combinations, including in combination with the right ventricular defibrillator coils, has not been performed. The researchers propose to investigate this method of optimisation.

A gold standard for optimisation of CRT has yet to be defined. Methods employed predominantly include invasive haemodynamic measurement and echocardiography. The ideal method would have low inter-observer variability, high ease of use and rapid sampling rate to allow adjustments to be made and evaluated quickly. USCOM, a continuous-wave Doppler method of continually assessing cardiac output, has been successfully used in optimisation of CRT and has gained a patent, however has so far been used to optimise atrio-ventricular delay only. This method may prove a more accurate, rapid and convenient way to rapidly assess response to changes in pacemaker parameters. The investigators plan to evaluate these three methods of assessment and correlate with each other and with cardiovascular outcomes.

Hypothesis:

Use of an algorithm in optimisation of cardiac resynchronisation therapy systems containing quadripolar left ventricular leads and dual coil right ventricular leads will increase response rate to this therapy.

Study structure:

Patients will be recruited consecutively amongst those undergoing implantation of a CRT-D device. At baseline, they will undergo assessment of functional capacity and echocardiographic parameters as well as invasive left ventricular pressure monitoring. The device will be implanted under normal laboratory conditions, aiming for a postero-lateral or lateral cardiac vein left ventricular lead position. Algorithmic echocardiography-guided optimisation of the devices will be conducted at the time of device implantation. Further assessment will be conducted simultaneously with haemodynamic left ventricular pressure monitoring and Ultrasound Cardiac Output Monitoring (USCOM) during device optimisation. The devices will then be programmed with standard CRT parameters. Subjects will be seen at 12 weeks for echocardiographic and functional assessment, following which algorithmic optimisation will be repeated with haemodynamic and echocardiographic monitoring concurrently. Further assessment will be performed at 24 weeks as per baseline, following which the study will end.

Study population: 24 men and women, 18 years and older, who are able to attend follow-up assessment 12 and 24 weeks after implantation.

ELIGIBILITY:
Inclusion Criteria:

* Successful implantation of CRT-D device with quadripolar left ventricular lead and dual coil right ventricular lead.

Exclusion Criteria:

* failed device implantation
* inability to complete the follow-up process
* inability to provide full written consent. Patients unable to perform cardiopulmonary exercise testing will be excluded from this assessment only and will be able to complete the remaining assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular end-systolic volume in patients undergoing algorithmic optimisation of CRT-D compared with usual device settings | 24 weeks
  End-systolic volume will be measured on echocardiography using Simpson's method. Where image quality precludes a full biplane assessment, single plane will be used with the apical 4-chamber view, or alternatively left ventricular end-systolic diameter will be used to calculate volume using the Teicholz method.

SECONDARY OUTCOMES:
Feasibility of algorithmic, echocardiography-guided CRT-D optimisation with quadripolar left ventricular leads in clinical practice | 24 weeks
  To see whether our optimisation algorithm is acceptable to patients and easy to perform in clinical practice.
Correlation between invasive haemodynamic studies with non-invasive ultrasound-based methods in optimising CRT-D | 24 weeks
  Attempt to establish a gold standard for optimisation of CRT devices by comparing invasive haemodynamic monitoring, echocardiographic parameters and cardiac output by ultrasound cardiac output monitoring (USCOM)
Change in left ventricular end diastolic pressure with algorithmic optimisation of CRT-D compared with usual device settings | 24 weeks
  A measurement of left ventricular end-diastolic pressure will be made via invasive left ventricular monitoring after programming with usual settings and again after programming using algorithmic optimisation of the CRT-D device.
Feasibility of ultrasound cardiac output monitoring (USCOM) in optimisation of CRT devices in clinical practice | At baseline and at 12 weeks
  Use of USCOM has been documented in optimisation of CRT, but not in such rapidly-changing algorithmic optimisation. We plan to assess whether it is feasible to use this in clinical practice as a replacement for a full echocardiogram.
Change in peak oxygen consumption with algorithmic CRT-D optimisation compared with usual device settings | 24 weeks
  Assessment of peak oxygen consumption as measured by cardiopulmonary exercise testing after usual settings compared with settings after algorithmic optimisation.
Change in left ventricular ejection fraction with algorithmic CRT-D optimisation compared with usual device settings. | 24 weeks
  Ejection fraction will be measured on echocardiography by Simpson's biplane method of discs. Where image quality precludes a full biplane assessment, single plane will be used with the apical 4-chamber view. Participants whose views are not sufficiently good quality for either of these measurements will be excluded from this outcome measure.
Change in left ventricular end-diastolic volume with algorithmic CRT-D optimisation compared with usual device settings. | 24 weeks
  End-diastolic volume will be measured on echocardiography using Simpson's method. Where image quality precludes a full biplane assessment, single plane will be used with the apical 4-chamber view, or the Teicholz method will be used to estimate end-diastolic volume by measuring left ventricular end-diastolic diameter.
Change in left ventricular diastolic filling time with algorithmic CRT-D optimisation compared with usual device settings. | 24 weeks
  Diastolic filling time will be measured on echocardiography using pulsed wave Doppler over the mitral inflow of the left ventricle.
Change in left ventricular outflow tract velocity time integral (LVOT VTI) with algorithmic CRT-D optimisation compared with usual device settings. | 24 weeks
  LVOT VTI will be measured on echocardiography using pulsed wave Doppler within the left ventricular outflow tract, within 1cm of the aortic valve where a clear envelope is visible.
Change in longitudinal and global longitudinal strain (GLS) with algorithmic CRT-D optimisation compared with usual device settings. | 24 weeks
  Longitudinal strain of the left ventricle will be measured on echocardiography using speckle tracking software
Change in radial strain with algorithmic CRT-D optimisation compared with usual device settings. | 24 weeks
  Radial strain of the left ventricle will be measured on echocardiography using speckle tracking software
Change in distance walked on a 6-minute hall walk test with algorithmic CRT-D optimisation compared with usual device settings | 24 weeks
  Patients will undergo a hall walk test at baseline, 12 weeks (with usual settings) and 24 weeks (following algorithmic optimisation) and the difference in distance walked will be analysed.
Change in New York Heart Association functional class with algorithmic CRT-D optimisation compared with usual device settings. | 24 weeks
  Functional status will be assessed at baseline, after 12 weeks (with usual settings) and after 24 weeks (with optimised settings) and the change in class will be recorded.
Change in score in the Minnesota Living with Heart Failure Questionnaire (MLHFQ) between algorithmically optimised CRT-D and usual device settings. | 24 weeks
  Patients will complete a questionnaire at baseline, 12 weeks (with usual settings) and 24 weeks (following algorithmic optimisation) and the difference in scores will be analysed. The Minnesota Living with Heart Failure Questionnaire is a validated and commonly used tool for assessing symptoms and activities of daily living in heart failure patients.
Change in cardiac output measured by the novel technique of Ultra-Sound Cardiac Output Monitoring (USCOM) with algorithmic CRT-D optimisation compared with usual device settings | 24 weeks
  USCOM is a validated technique that correlates well with echocardiographic and Doppler measurements of cardiac output and is performed using a simple probe placed at several points over the chest wall.
Number of patients suffering adverse events during the study period | From patient enrollment through study completion, an average of 1 year.
  Hospital patient record systems and telephone calls will be used to find out about hospital admissions and mortality during the study period. An adverse event will be defined as an admission to hospital or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Freya M Lodge, MBBS, Principal Investigator — Cardiff and Vale University Health Board; Zaheer R Yousef, MBBS, Study Director — Cardiff and Vale University Health Board
Locations (1):
- University Hospital of Wales, Cardiff, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data available on individual written request at the discretion of the investigators.

REFERENCES:
- [Background] Auricchio A, Stellbrink C, Sack S, Block M, Vogt J, Bakker P, Huth C, Schondube F, Wolfhard U, Bocker D, Krahnefeld O, Kirkels H; Pacing Therapies in Congestive Heart Failure (PATH-CHF) Study Group. Long-term clinical effect of hemodynamically optimized cardiac resynchronization therapy in patients with heart failure and ventricular conduction delay. J Am Coll Cardiol. 2002 Jun 19;39(12):2026-33. doi: 10.1016/s0735-1097(02)01895-8. PMID 12084604
- [Background] Abraham WT, Fisher WG, Smith AL, Delurgio DB, Leon AR, Loh E, Kocovic DZ, Packer M, Clavell AL, Hayes DL, Ellestad M, Trupp RJ, Underwood J, Pickering F, Truex C, McAtee P, Messenger J; MIRACLE Study Group. Multicenter InSync Randomized Clinical Evaluation. Cardiac resynchronization in chronic heart failure. N Engl J Med. 2002 Jun 13;346(24):1845-53. doi: 10.1056/NEJMoa013168. PMID 12063368
- [Background] Young JB, Abraham WT, Smith AL, Leon AR, Lieberman R, Wilkoff B, Canby RC, Schroeder JS, Liem LB, Hall S, Wheelan K; Multicenter InSync ICD Randomized Clinical Evaluation (MIRACLE ICD) Trial Investigators. Combined cardiac resynchronization and implantable cardioversion defibrillation in advanced chronic heart failure: the MIRACLE ICD Trial. JAMA. 2003 May 28;289(20):2685-94. doi: 10.1001/jama.289.20.2685. PMID 12771115
- [Background] Daubert C, Gold MR, Abraham WT, Ghio S, Hassager C, Goode G, Szili-Torok T, Linde C; REVERSE Study Group. Prevention of disease progression by cardiac resynchronization therapy in patients with asymptomatic or mildly symptomatic left ventricular dysfunction: insights from the European cohort of the REVERSE (Resynchronization Reverses Remodeling in Systolic Left Ventricular Dysfunction) trial. J Am Coll Cardiol. 2009 Nov 10;54(20):1837-46. doi: 10.1016/j.jacc.2009.08.011. Epub 2009 Oct 1. PMID 19800193
- [Background] Linde C, Abraham WT, Gold MR, St John Sutton M, Ghio S, Daubert C; REVERSE (REsynchronization reVErses Remodeling in Systolic left vEntricular dysfunction) Study Group. Randomized trial of cardiac resynchronization in mildly symptomatic heart failure patients and in asymptomatic patients with left ventricular dysfunction and previous heart failure symptoms. J Am Coll Cardiol. 2008 Dec 2;52(23):1834-1843. doi: 10.1016/j.jacc.2008.08.027. Epub 2008 Nov 7. PMID 19038680
- [Background] Chung ES, Katra RP, Ghio S, Bax J, Gerritse B, Hilpisch K, Peterson BJ, Feldman DS, Abraham WT. Cardiac resynchronization therapy may benefit patients with left ventricular ejection fraction >35%: a PROSPECT trial substudy. Eur J Heart Fail. 2010 Jun;12(6):581-7. doi: 10.1093/eurjhf/hfq009. Epub 2010 Feb 11. PMID 20150328
- [Background] Osca J, Alonso P, Cano O, Andres A, Miro V, Tello MJ, Olague J, Martinez L, Salvador A. The use of multisite left ventricular pacing via quadripolar lead improves acute haemodynamics and mechanical dyssynchrony assessed by radial strain speckle tracking: initial results. Europace. 2016 Apr;18(4):560-7. doi: 10.1093/europace/euv211. Epub 2015 Sep 1. PMID 26333378
- [Background] Rinaldi CA, Burri H, Thibault B, Curnis A, Rao A, Gras D, Sperzel J, Singh JP, Biffi M, Bordachar P, Leclercq C. A review of multisite pacing to achieve cardiac resynchronization therapy. Europace. 2015 Jan;17(1):7-17. doi: 10.1093/europace/euu197. Epub 2014 Sep 11. PMID 25214507
- [Background] Pappone C, Calovic Z, Vicedomini G, Cuko A, McSpadden LC, Ryu K, Romano E, Saviano M, Baldi M, Pappone A, Ciaccio C, Giannelli L, Ionescu B, Petretta A, Vitale R, Fundaliotis A, Tavazzi L, Santinelli V. Multipoint left ventricular pacing improves acute hemodynamic response assessed with pressure-volume loops in cardiac resynchronization therapy patients. Heart Rhythm. 2014 Mar;11(3):394-401. doi: 10.1016/j.hrthm.2013.11.023. Epub 2013 Nov 28. PMID 24291411
- [Background] Siu CW, Tse HF, Lee K, Chan HW, Chen WH, Yung C, Lee S, Lau CP. Cardiac resynchronization therapy optimization by ultrasonic cardiac output monitoring (USCOM) device. Pacing Clin Electrophysiol. 2007 Jan;30(1):50-5. doi: 10.1111/j.1540-8159.2007.00579.x. PMID 17241315
- [Background] Zanon F, Baracca E, Pastore G, Marcantoni L, Fraccaro C, Lanza D, Picariello C, Aggio S, Roncon L, Dell'Avvocata F, Rigatelli G, Pacetta D, Noventa F, Prinzen FW. Multipoint pacing by a left ventricular quadripolar lead improves the acute hemodynamic response to CRT compared with conventional biventricular pacing at any site. Heart Rhythm. 2015 May;12(5):975-81. doi: 10.1016/j.hrthm.2015.01.034. Epub 2015 Jan 24. PMID 25625721